CLINICAL TRIAL: NCT03151733
Title: Single Incision Laparoscopic Surgery (SILS) for Colorectal Disease
Brief Title: Single Incision Laparoscopic Colorectal Surgery
Acronym: SILCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Ren, chief physicion, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJ-SILS-CRC2017; SHSDC (Other: SHSDC)
Record Dates: First submitted 2017-03-20; First posted 2017-05-12 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Laparoscopic Colorectal Surgery
Keywords: SILS; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single incision laparoscopic surgery (Experimental): patients with colorectal cancer and undergo single incision laparoscopic surgery
  Interventions: Procedure: single incision laparoscopic surgery
- Conventional laparoscopic surgery (Placebo Comparator): patients with colorectal cancer and undergo conventional laparoscopic surgery
  Interventions: Procedure: conventional laparoscopic surgery

INTERVENTIONS:
Procedure: single incision laparoscopic surgery — Patients undergo single incision laparoscopic surgery
  Arms: single incision laparoscopic surgery
Procedure: conventional laparoscopic surgery — Patients undergo conventional laparoscopic surgery
  Arms: Conventional laparoscopic surgery

SUMMARY:
Single incision laparoscopic surgery (SILS) is the further development of the concept of minimally invasive surgery for colorectal cancer,which rapidly developed in the field of colorectal surgery. Through the development of single hole laparoscopic colorectal cancer radical surgery and clinical study and follow up accordingly, evaluating the feasibility, surgical effectiveness and economy help to promote the popularization and application of single hole laparoscopic techniques in the field.

DETAILED DESCRIPTION:
The patients with colorectal cancer will randomly divided into single incision laparoscopic surgery group and conditional laparoscopic surgery group. The operation time, blood loss, the incidence of lymph node , the number of postoperative complications, the gastrointestinal function recovery time, postoperative hospital stay，the number of local recurrence and distant metastasis, survival rate and the total cost of hospitalization will be evaluated to confirm the feasibility of single incision laparoscopic surgery is effective and economical. It is worthy of clinical application.

ELIGIBILITY:
Inclusion Criteria:

* 18 years < age < 80 years
* Tumor located in colon and high rectum ( the lower border of the tumor is above the peritoneal reflection)
* Pathological colorectal carcinoma
* Clinically diagnosed cT1-4aN0-2 M0 lesions according to the 7th Edition of AJCC Cancer Staging Manual
* Tumor size of 5 cm or less
* ECOG score is 0-1
* ASA score is Ⅰ-Ⅲ
* Informed consent

Exclusion Criteria:

* Body mass index (BMI) >30 kg/m2
* The lower border of the tumor is located distal to the peritoneal reflection
* Pregnant woman or lactating woman
* Severe mental disease
* Previous abdominal surgery（except appendectomy and cholecystotomy）
* Emergency operation due to complication (bleeding, perforation or obstruction) caused by colorectal cancer
* Requirement of simultaneous surgery for other disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2019-06-29 (Actual); Study Completion 2024-06-29 (Actual)

PRIMARY OUTCOMES:
Early morbidity rate | 30 days
  morbidity rate 30 days after surgery

SECONDARY OUTCOMES:
Operative time | intraoperative
  Operative time（minutes）
Intraoperative blood loss | intraoperative
  Estimated blood loss（milliliters，ml）
Incision length | intraoperative
  Incision length（centimeters，cm）
Lymph node detection | 14 days after surgery
  Lymph nodes harvested（numbers）
Incisal margin | 14 days after surgery
  Length of proximal and distal margin （centimeters，cm）
Tumor size | 14 days after surgery
  The diameter of tumors（centimeters，cm）
Length of stay | 1-14 days after surgery
  Duration of hospital stay（days after surgery）
Postoperative recovery course | 1-14 days after surgery
  Time to first ambulation, flatus, liquid diet and soft diet （hours after surgery）
Pain score | 1-3 days after surgery
  Postoperative pain is recorded using the visual analog scale (VAS) pain score （0-10 points）tool on postoperative day 1, 2, 3 and the day of discharge
3-year disease free survival rate | 36 months after surgery
  3-year disease free survival rate
5-year overall survival rate | 60 months after surgery
  5-year overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Liu Kun, MD, Study Chair — ruijin hospitla North
Locations (1):
- ruijin hospital North, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aldeghaither S, Zubaidi A, Alkhayal K, Al-Obaid O. Single-incision laparoscopic colorectal surgery: a report of 33 cases in Saudi Arabia. Ann Saudi Med. 2016 Jul-Aug;36(4):282-7. doi: 10.5144/0256-4947.2016.282. PMID 27478914
- [Derived] Song Z, Liu K, Li Y, Shi Y, Jiang Y, Wang C, Chen X, Zhang T, Ji X, Zhao R. Short-Term Outcomes of Single-Incision Laparoscopic Surgery for Colorectal Cancer: A Single-Center, Open-Label, Non-Inferiority, Randomized Clinical Trial. Front Oncol. 2021 Oct 25;11:762147. doi: 10.3389/fonc.2021.762147. eCollection 2021. PMID 34760706
- [Derived] Song Z, Li Y, Liu K, Jiang Y, Shi Y, Ji X, Zhang T, Wu H, Shi Y, Zhao R. Clinical and oncologic outcomes of single-incision laparoscopic surgery for right colon cancer: a propensity score matching analysis. Surg Endosc. 2019 Apr;33(4):1117-1123. doi: 10.1007/s00464-018-6370-2. Epub 2018 Jul 24. PMID 30043168